CLINICAL TRIAL: NCT03734848
Title: Bilateral Ultrasound Guided Pectoralis Nerve Block Induces Hemodynamic Stability With Reducing Systemic Stress Response for Adult Patients Undergoing Off-pump Coronary Artery Bypass Graft
Brief Title: Bilateral Ultrasound Guided Pectoralis Nerve Block Induces Hemodynamic Stability With Reducing Systemic Stress Response for Off-pump Coronary Artery Bypass Graft
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Said Elgebaly,MD, director, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TantaS
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Analgesic Effects; Systemic Stress Response; Hemodynamic Stability
Keywords: Pectoralis block; Opioids Consumption; off-pump

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (No Intervention): patients did not receive Bilateral Ultrasound Guided Pectoralis Nerve Block (control group).
- Group 2 (Active Comparator): patients receive Bilateral Ultrasound Guided Pectoralis Nerve Block (control group).
  Interventions: Drug: Bilateral Ultrasound Guided Pectoralis Nerve Block.

INTERVENTIONS:
Drug: Bilateral Ultrasound Guided Pectoralis Nerve Block. — Using a 20-gauge 5 cm needle. Injection bupivacaine 0.25% used as a local anesthetic. The block was performed in a supine position with the arm slightly abducted. The ultrasound probe was placed at the midclavicular level infero-laterally to locate the axillary artery and vein and then moved laterally toward the axilla until pectoralis major, pectoralis minor, and serratus anterior muscles were identified at the level of the fourth rib. The needle was inserted in-plane with respect to the ultrasound probe. A volume of 20 ml of local anesthetic solution was deposited in the fascial plane between pectoralis minor and serratus anterior muscle, followed by withdrawal of the needle to the fascial plane between the pectoralis major and pectoralis minor muscle, where a volume of 10 ml was deposited. The block was performed similarly on the opposite side. Care was taken not to cross the toxic dose of bupivacaine (3 mg/kg).
  Arms: Group 2

SUMMARY:
Opioids used in attenuation of the neuroendocrine stress response in patients undergoing off-pump coronary artery bypass graft (OPCAB) it produces predictable satisfactory analgesia and sedation but with side effects such as respiratory depression, drowsiness, and myocardial depression. Regional techniques may be encouraged to be anti-stress procedures and produce risk-free postoperative (OPCAB) period. Pectoralis nerve block (pecs block) appears to possess a great deal of promise for patients undergoing (OPCAB) because of low complication rates as it is less invasive regional analgesic technique when compared to paravertebral, thoracic epidural analgesia and parenteral analgesia.

DETAILED DESCRIPTION:
Aims: Ultrasound Guided Bilateral Pecs block would provide attenuation of the neuroendocrine stress response with hemodynamic profile stability, decreased analgesic consumption and improves patient postoperative outcomes after(OPCAB).

Materials and Methods: A prospective, single-blind, controlled study enrolled forty patients between the age groups of 25 and 65 years undergoing (OPCAB) through midline sternotomy under general anesthesia and randomly allocated into two groups with 20 in each group. Group 1 patients did not receive Pecs block (control group), patients were anesthetized to keep the heart rate and blood pressure within 25% of the baseline values. Whereas Group 2 patients received bilateral Pecs block preoperatively. Patients were extubated once they fulfilled extubation criteria. Heart rate, mean arterial blood pressure, Plasma levels of adrenocorticotropic hormone(ACTH) and cortisol, sufentanil consumption were determined at the following points: Basically (T0),immediately before the induction of anesthesia; (T1), immediately after tracheal intubation; (T2),immediately after sternotomy;( T3), 30 minutes after the start of surgery; and (T4), at the end of surgery. Ventilator duration, duration of ICU stay hospital stay were recorded postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing first-time OPCAB surgery.
* patients with good or only slightly reduced left ventricular function (ejection fraction _40%, left ventricular end-diastolic pressure _15 mmHg)
* patients below 75years of age

Exclusion Criteria:

* patients requiring CPB either electively or during the course of surgery
* patients with renal insufficiency (creatinine _1.5 mg/dL) or hepatic impairment (alanine aminotransferase or aspartate aminotransferase _40 U/mL)
* patients who misused alcohol or drugs
* patients with hemodynamic instability
* symptoms of congestive cardiac failure
* preexisting infection at the block site
* allergy to local anesthetics
* psychiatric illness
* patients with prolonged postoperative ventilator course

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Changes in Heart rate. | Basically (T0),immediately before the induction of anesthesia; (T1), immediately after tracheal intubation; (T2),immediately after sternotomy;( T3), 30 minutes after the start of surgery; and (T4), immediately at the end of surgery
  Ranges of heart rate will be estimated in beat per minutes.
changes in mean arterial blood pressure and cardiac indices. | Basically (T0),immediately before the induction of anesthesia; (T1), immediately after tracheal intubation; (T2),immediately after sternotomy;( T3), 30 minutes after the start of surgery; and (T4),immediately at the end of surgery
  Ranges of mean arterial blood pressure estimated in mmHg.
changes in cardiac indices. | Basically (T0),immediately before the induction of anesthesia; (T1), immediately after tracheal intubation; (T2),immediately after sternotomy;( T3), 30 minutes after the start of surgery; and (T4),immediately at the end of surgery
  Ranges of Cardiac indices will be estimated as follow :CO in (L/min),Cl in (L/min/m2),SVR in (dyn•s/cm5) and PVR in (dyn•s/cm5).
changes in Plasma levels of adrenocorticotropic hormone(ACTH) . | Basically (T0),immediately before the induction of anesthesia; (T1), immediately after tracheal intubation; (T2),immediately after sternotomy;( T3), 30 minutes after the start of surgery; and (T4),immediately at the end of surgery
  Ranges in Plasma levels of adrenocorticotropic hormone(ACTH) in (pg/mL) and cortiso in l(ng/mL)
changes in Plasma levels of cortisol hormone | Basically (T0),immediately before the induction of anesthesia; (T1), immediately after tracheal intubation; (T2),immediately after sternotomy;( T3), 30 minutes after the start of surgery; and (T4), immediately at the end of surgery
  Ranges in Plasma levels of cortisol in (ng/mL)

SECONDARY OUTCOMES:
changes in sufentanil consumption | Basically (T0),immediately before the induction of anesthesia; (T1), immediately after tracheal intubation; (T2),immediately after sternotomy;( T3), 30 minutes after the start of surgery; and (T4),immediately at the end of surgery
  Measured by (µg/kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Said Elgebaly, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kumar KN, Kalyane RN, Singh NG, Nagaraja PS, Krishna M, Babu B, Varadaraju R, Sathish N, Manjunatha N. Efficacy of bilateral pectoralis nerve block for ultrafast tracking and postoperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):333-338. doi: 10.4103/aca.ACA_15_18. PMID 30052231
- [Result] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Result] Froyshteter AB, Bhalla T, Tobias JD, Cambier GS, Mckee CT. Pectoralis blocks for insertion of an implantable cardioverter defibrillator in two patients with Duchenne muscular dystrophy. Saudi J Anaesth. 2018 Apr-Jun;12(2):324-327. doi: 10.4103/sja.SJA_624_17. PMID 29628849
- [Result] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533